CLINICAL TRIAL: NCT02049268
Title: Neural Mechanisms Underlying Nicotine and Alcohol Combinations
Acronym: QfMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Lisa Nickerson, PhD, Instructor in Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012P000217
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Focus: Effects of Nicotine and Alcohol on Brain Circuits
Keywords: alcohol; nicotine; addiction; functional MRI; functional connectivity; brain circuits
MeSH Terms: conditions — Behavior, Addictive | interventions — Nicotine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nicotine + Alcohol (Experimental): A nicotine patch will be applied to the subject. After a 3-4 hour uptake period, subjects will undergo a single MRI session. Baseline (nicotine only) measurements will be made, then participants will drink an alcoholic beverage. Post-alcohol measurements will be made after a 20 minute uptake period.
  Interventions: Drug: Nicotine + Alcohol
- Placebo Nicotine + Alcohol (Experimental): A placebo nicotine patch will be applied to the subject. After a 3-4 hour uptake period, subjects will undergo a single MRI session. Baseline (placebo nicotine) measurements will be made, then participants will drink an alcoholic beverage. Post-alcohol measurements will be made after a 20 minute uptake period.
  Interventions: Drug: Placebo Nicotine + Alcohol
- Nicotine + Placebo Alcohol (Experimental): A nicotine patch will be applied to the subject. After a 3-4 hour uptake period, subjects will undergo a single MRI session. Baseline (nicotine only) measurements will be made, then participants will drink a placebo alcoholic beverage. Post-alcohol measurements will be made after a 20 minute uptake period.
  Interventions: Drug: Nicotine + Placebo Alcohol

INTERVENTIONS:
Drug: Nicotine + Alcohol — 14 mg nicotine patch applied in combination with vodka and orange juice alcoholic beverage (to reach blood alcohol level (BAL) = 0.08 based on subject weight, which is approximately 2-3 drinks for 400 mL volume)
  Other Names: Nicoderm CQ Clear; Absolute Vodka
  Arms: Nicotine + Alcohol
Drug: Placebo Nicotine + Alcohol — Placebo nicotine patch applied in combination with vodka and orange juice alcoholic beverage (to reach BAL = 0.08 based on subject weight, which is approximately 2-3 drinks for 400 mL volume)
  Other Names: Nicoderm CQ Clear; Absolute Vodka
  Arms: Placebo Nicotine + Alcohol
Drug: Nicotine + Placebo Alcohol — 14 mg nicotine patch applied in combination with 400 mL orange juice beverage with a trace of alcohol to create placebo alcohol mixture.
  Other Names: Nicoderm CQ Clear; Absolute Vodka
  Arms: Nicotine + Placebo Alcohol

SUMMARY:
Nicotine and alcohol are frequently used together and their combined use contributes to more than half a million deaths each year, with more alcoholics dying from smoking-related diseases than from alcohol-related diseases. Using a new multi-modal MRI approach combined with data fusion, the investigators propose to study how nicotine modulates alcohol-induced changes in the function of brain circuits. The investigators hypotheses are:

* functional connectivity (FC) in the reward network, containing components of the mesolimbic dopamine system, will be altered by alcohol, and additional increases in FC will be observed if nicotine is also present (e.g., additive effects).
* co-administration of nicotine will counteract the effects of alcohol on FC in multiple brain networks, including visual, sensorimotor and motor brain circuits, that may be associated with the impairing effects of alcohol

DETAILED DESCRIPTION:
Long-term Objectives: Our long-term objective is to bring together non-invasive quantitative functional magnetic resonance imaging (q-fMRI) with a newly developed cutting-edge analysis method to study changes in neuronal metabolism and cerebrovascular function that occurs during psychoactive drug use.

Specific Aims: Our first specific aim is to validate the components of the q-fMRI acquisition, which requires several different kinds of fMRI scans (or multimodal measurements). The second aim then applies the q-MRI method to study the functional brain networks that define brain activity when a person is simply resting and not engaged in any activity. These networks each consist of a unique set of regions that spontaneously fluctuate together in order to be "tuned" for future task performance. The effects of nicotine and alcohol and their interaction on these resting state networks are the focus of the application of our new q-fMRI strategy. q-fMRI measurements require several different scans, including making measurements of perfusion and oxygen metabolism, and an integrated analysis of all of these different results will be much more informative than separate analyses of each measurement. However, the analysis method, the linked independent component analysis (linked ICA) approach is very new and has never been applied to q-fMRI measurements or any other measurements of psychoactive drug effects. Thus, the third aim is to apply this novel analysis method to data acquired under different drug conditions to identify patterns of related activity in our multimodal fMRI data.

Research Design and Methods: A randomized within-subject study of 23 healthy subjects will be done as follows: fMRI scanning will begin four hours after pre-treatment with either nicotine or placebo patch (randomized). Alcohol will then be consumed by subjects while in the scanner and a second scanning session will be done of the combination of nicotine (placebo) + alcohol to assess changes in resting state functional connectivity due to alcohol and nicotine and their interactions.

Significance: Linked ICA with q-fMRI measurements is an innovative strategy for studying brain function that could have a significant impact in the ability of fMRI to give an integrated picture of the spectrum of effects that drugs of abuse may have on brain function, and is thus ideally suited to the goals of the CEBRA mechanism. By applying this technique to study alcohol and nicotine co-use, we also will contribute greatly to the understanding of this significant health problem.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 21 to 40 years old
* Physically healthy (normal physical exam, ECG, blood and urine chemistries)
* Light/moderate cigarette smokers (greater than 10-20 cigarettes per week)
* Alcohol drinkers (10 or greater drinks per week)
* Must not be seeking treatment for their alcohol or tobacco use

Exclusion Criteria:

* Female
* Diagnosis of past or current alcohol dependence as assessed by Diagnostic and Statistic Manual, DSM-IV, criteria for alcohol dependence
* Diagnosis of cocaine, sedative, or opiate dependence using DSM-IV criteria
* Current diagnosis of Axis I disorder using DSM-IV criteria, or any Axis I disorder within past 5 years (excluding alcohol abuse, marijuana dependence or abuse)
* Current daily use of antipsychotic, antidepressant, or other psychoactive prescription drug, as well as daily use of non-prescription drugs
* Life threatening or unstable medical illness, or one that can create marked change in mental state
* Heavy caffeine use (greater than 400 mg on a regular, daily basis)
* History of seizure disorder
* Hepatitis B or C positive, or history of i.v. drug use

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functional connectivity of reward-related brain circuit | 1.5 hours
  In a single 1.5 hour MRI session, functional connectivity of the reward circuit will be assessed with either nicotine or placebo nicotine on board. Participants will then drink an alcoholic or placebo alcohol beverage (whilst still in the scanner) and will be rescanned after a 20 minute resting period (also still in the scanner). The primary outcome is the pre- minus the post-alcohol functional connectivity of the reward brain circuit.

SECONDARY OUTCOMES:
Exploratory investigation of oxygen metabolism and perfusion underlying the functional connectivity effects | 1.5 hours
  An exploratory data fusion approach will be applied to the MRI measurements to evaluate patterns of related cerebrovascular and neural function in all brain circuits that are associated with nicotine and alcohol effects.
Functional connectivity of visual, motor, and sensorimotor brain circuits | 1.5 hours
  In a single 1.5 hour MRI session, functional connectivity of the reward circuit will be assessed with either nicotine or placebo nicotine on board. Participants will then drink an alcohol or placebo alcohol beverage (whilst still in the scanner) and will be rescanned after a 20 minute resting period (also still in the scanner). The primary outcome is the pre- minus the post-alcohol functional connectivity for each brain circuit.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Nickerson, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing will be considered on a case by case basis to ensure IRB compliance.